CLINICAL TRIAL: NCT05695976
Title: A Study for Patients Newly Diagnosed With Glioblastoma Being Treated With Standard Radiotherapy and Temozolomide (TMZ) to Evaluate Tumor Response Via Liquid Biopsies (GRETeL)
Brief Title: GRETeL: Tumor Response to Standard Radiotherapy and TMZ Patients With GBM
Status: Suspended | Type: Observational
Why Stopped: The study is suspended while preplanned interim analysis is being completed.
Sponsor: Duke University (Other)
Collaborators: Personalis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00110247
Record Dates: First submitted 2022-12-20; First posted 2023-01-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma; Glioma, Malignant
Keywords: Khasraw; Glioblastoma; Glioma; Pro00110247; GRETEL; Duke
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor (archival) specimens will be obtained from the surgical resection and diagnosis of GBM and before initiation of radiotherapy. It is anticipated that a certain proportion of patients will need to undergo further tumor debulking after radiotherapy. In such instances, these post-radiotherapy re-resected tumor specimens will also be collected for later sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilot: The first 20 patients accrued to this study will be assayed to validate the performance of the assays developed by Personalis. This pilot sub-study will be analyzed in a "blinded" manner without clinical information.
- Full Study: The remaining 80 patients accrued to this study (after the initial 20 patients accrue to the "Pilot" cohort).

SUMMARY:
The purpose of this study is to better define longitudinal genomic alterations in patients with glioblastoma (GBM), and to determine if plasma circulating tumor DNA (ctDNA) or cell free DNA (cfDNA) is associated with disease recurrence, survival, tumor characteristics, and/or peripheral immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients newly diagnosed with malignant glioma, IDH wildtype who have undergone surgical resection for their tumor and who are planned for standard of care radiation therapy with concurrent temozolomide (i.e., at least 59 Gy in 30 fractions over 6 weeks)
* Patients must have leftover tissue available from the surgical resection of their tumor available to request for this research.
* Able to undergo MRI of brain with and without contrast
* Signed informed consent approved by the Institutional Review Board (IRB)

Exclusion Criteria:

* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with glioblastoma post-resection who are scheduled to receive standard radiation and chemotherapy (temozolomide).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Median cf/ctDNA concentration at pre- and post-radiation, as well as median change in ct/ctDNA concentration | 6 months
  Identify and describe changes in the cell free DNA (cfDNA) sequencing profiles of patients diagnosed with GBM in pre- versus post-radiation therapy samples, and to assess the association between these changes and clinical outcome, including progression free and overall survival
Median levels of cfDNA collected longitudinally after completion of radiation | 6 months
  Identify and describe changes over time after radiotherapy in the cfDNA sequencing profiles of patients diagnosed with GBM, and to assess the association between these longitudinal changes in cfDNA and clinical outcome, including progression free and overall survival

OTHER OUTCOMES:
Characterize the fragmentomic landscape of GBM | 6 months
  Median number of ctDNA fragments obtained from tumor tissue, pre-radiation serum specimen, and post-radiation serum specimen, and healthy controls.
Spearman correlation between clinical descriptors and measures of ctDNA | 6 months
  Assess the association between degree and frequency of ctDNA shedding and clinical characteristics, such as molecular findings, histopathological characteristics, corticosteroid use, and bevacizumab use.
Median and range for measures of tumor immune infiltration | 6 months
  Quantify the level of immune infiltration in the tumor, and assess its association with progression-free survival (PFS), overall survival (OS), and ctDNA detection.
Hazard ratio for the relationship between chromosomal instability and OS or PFS | 6 months
  Assess the prognostic value of chromosomal instability/CAN burden, and assess its association with ctDNA from plasma.
Spearman correlation between ctDNA and peripheral T cell function, autoantibodies. | 6 months
  Determine if peripheral T cell function and stemness or autoantibodies are association with ctDNA levels, or TME composition.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Center at Duke University — http://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://www.dukehealth.org/clinical-trials